CLINICAL TRIAL: NCT04243421
Title: Clinical and Radiographic Evaluation of the Marginal Bone and Soft Tissue Alterations After the Treatment With Use of OsseoSpeed EV Profile Implants: A Case Series Study
Brief Title: Marginal Bone and Soft Tissue Alterations After Use of OsseoSpeed EV Profile Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry); Dental Practice, Malgorzata Pietruska, Jan Pietruski (Other)
Responsible Party: Principal Investigator, Małgorzata Pietruska, professor, Medical University of Bialystok
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N/ST/ZB/18/001/1164; D-2013-010 (Other Grant/Funding Number: Dentsply Sirona Implants)
Record Dates: First submitted 2020-01-18; First posted 2020-01-28 (Actual); Results first posted 2021-01-13 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Alveolar Process Atrophy
Keywords: implant; soft tissue
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: case series
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group with implants (Experimental): Flap will be elevated following the crestal and releasing incisions (if necessary).
  After having completed the cleaning, the surgeon will perform the osteotomy. After the use of the final drill ᴓ3.2 the surgeon will take the measurement of the buccal and palatal/lingual walls height.
  If wall discrepancy is 1.5-2mm the site will be included in the study. Clinical photographs of probe within the osteotomy have to be taken. The osteotomy will be prepared with the conical drill, therefore the implant will be inserted in a special manner - lower part of the sloped collar will be located at the buccal aspect of the osteotomy preparation. At the buccal aspect the implant will positioned at the crestal bone level, while at the palatal aspect it will be either at the level of the bone crest or 0.5 mm below.
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Soft tissue aesthetics, marginal bone level on CBCT

SUMMARY:
Evaluation of the marginal bone and soft tissue alterations after the OsseoSpeed™ EV Profile implants placement in anterior maxilla.

The following parameters will be tested:

* pink esthetic score - at the temporary crown delivery, at the final crown delivery, 6 months post final crown delivery
* papilla index - at the temporary crown delivery, at the final crown delivery, 6 months post final crown delivery
* changes in radiographic marginal bone levels and width at buccal and palatal aspects: differences between baseline (the day of surgery) and 1-year post-op measurements on CBCT will be made.

DETAILED DESCRIPTION:
Surgical procedures

Flap will be elevated following the crestal and releasing incisions (if necessary).

After having completed the cleaning, the surgeon will perform the osteotomy. After the use of the final drill ᴓ3.2 the surgeon will take the measurement of the buccal and palatal/lingual walls height.

If wall discrepancy is 1.5-2mm the site will be included in the study. Clinical photographs of probe within the osteotomy have to be taken. The osteotomy will be prepared with the conical drill, therefore the implant will be inserted in a special manner - lower part of the sloped collar will be located at the buccal aspect of the osteotomy preparation. At the buccal aspect the implant will positioned at the crestal bone level, while at the palatal aspect it will be either at the level of the bone crest or 0.5 mm below.

The flap will be sutured with 5/0 or 6/0 non-absorbable Ethilon sutures using the mattress and single interrupted sutures. Clinical photographs of the treated site after flap suturing will be taken.

Post-surgical instructions and follow-up

* Ibuprofen 400 mg 2-4 times per day will be prescribed in case of pain. In case of gastric problems it will be replaced by Paracetamol 1 g (max 4 g per day).
* Patient will be reminded to go on with the antibiotic prophylactic therapy as previously described.
* Chlorhexidine mouthwash 0.12% for 1 minute twice a day for 3 weeks will be provided.
* Suture removal after 2 weeks.

Check-ups and maintenance Appointments will be scheduled at weeks 1, 2, 4, and 6. Clinical photographs will be taken. During these appointments the presence of suppuration and flap dehiscence will be recorded dichotomously as presence/absence.

Uncovering procedure will be scheduled at 8 weeks post-op. After crestal incision and gentle flap elevation the height of denudated buccal implant surface (if present) will be measured using a periodontal probe. Then the healing abutment will be screwed in and single interrupted sutures will be placed with the use 5/0 or 6/0 non-absorbable Ethilon sutures (if necessary). Suture removal is planned 7 days after procedure. Clinical photographs will be taken.

Temporary crown will be delivered 3 months post implant placement. Clinical examination (PES, PI) will be performed. Photographs and control CBCT will be taken.

Final prosthetic reconstruction will be delivered 6 months post-op. Clinical examination (PES, PI) will be performed as well as clinical photographs will be taken.

1 year evaluation Clinical examination (PES, PI) will be performed. Clinical photographs of the study site will be taken. Control CBCT will be taken.

In case of any complication observed during any of the scheduled visit or during an emergency visit, intraoral radiographs and clinical photographs will be taken and the CRF will be filled in.

ELIGIBILITY:
Inclusion Criteria:

* lack of tooth in position of central incisors, canines and premolars

Exclusion Criteria:

* Smoking
* Uncontrolled diabetes
* Pregnancy or lactation
* Poor oral hygiene
* Compromised dentition neighboring to edentulous site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pietruski, Study Chair — Praktyka Stomatologiczna M. J. Pietruscy
Locations (1):
- Małgorzata Pietruska, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemt T. Regeneration of gingival papillae after single-implant treatment. Int J Periodontics Restorative Dent. 1997 Aug;17(4):326-33. PMID 9497723
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100

RESULTS

PARTICIPANT FLOW:
Groups:
- Group With Implants: Flap will be elevated following the crestal and releasing incisions (if necessary).
  After having completed the cleaning, the surgeon will perform the osteotomy. After the use of the final drill ᴓ3.2 the surgeon will take the measurement of the buccal and palatal/lingual walls height.
  If wall discrepancy is 1.5-2mm the site will be included in the study. Clinical photographs of probe within the osteotomy have to be taken. The osteotomy will be prepared with the conical drill, therefore the implant will be inserted in a special manner - lower part of the sloped collar will be located at the buccal aspect of the osteotomy preparation. At the buccal aspect the implant will positioned at the crestal bone level, while at the palatal aspect it will be either at the level of the bone crest or 0.5 mm below.
  Implantation: Soft tissue aesthetics, marginal bone level on Cone Beam Computed Tomography (CBCT).
Period: Overall Study
Arm/Group | Group With Implants
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group With Implants: Flap will be elevated following the crestal and releasing incisions (if necessary).
  After having completed the cleaning, the surgeon will perform the osteotomy. After the use of the final drill ᴓ3.2 the surgeon will take the measurement of the buccal and palatal/lingual walls height.
  If wall discrepancy is 1.5-2mm the site will be included in the study. Clinical photographs of probe within the osteotomy have to be taken. The osteotomy will be prepared with the conical drill, therefore the implant will be inserted in a special manner - lower part of the sloped collar will be located at the buccal aspect of the osteotomy preparation. At the buccal aspect the implant will positioned at the crestal bone level, while at the palatal aspect it will be either at the level of the bone crest or 0.5 mm below.
  Implantation: Soft tissue aesthetics, marginal bone level on CBCT
Arm/Group | Group With Implants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 30

OUTCOME MEASURES:

1. Primary Outcome: Pink Esthetic Score (PES) at Temporary Crown Delivery.
Description: Pink Esthetic Score (PES): 0-10; minimum - 0, maximum - 10; the best outcome: 10 PES subscores: mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, root convexity/soft tissue color and texture at the facial aspect of the implant site. Minimum 0, maximum - 2; the best outcome: 2
Time Frame: value changes between examination carried out 3 and 9 months post-op
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group With Implants
Number analyzed (Participants) | 30
score on a scale
  Mesial papilla | 1 [0 to 1]
  Distal papilla | 1 [0 to 1]
  Curvature of the facial mucosa | 1 [0.5 to 2]
  Level of the facial mucosa | 1 [0.5 to 2]
  Root convexity/soft tissue color and texture | 1 [1 to 2]
  Pink Esthetic Score | 5 [3 to 8]
Statistical Analysis 1: Comparison: Group With Implants; Test type: Other; p = 0.0007, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 6

2. Primary Outcome: Papilla Index (PI) at Temporary Crown Delivery.
Description: Papilla Index score: 0-4; the best outcome: 3; minimum: 0, maximum: 4 0 - no papilla present; 1 - less than half of the height of papilla present; 2 - half or more of the height of papilla is present but does not extend all the way up to the contact point between of the crowns; 3 - the papilla fill up the entire proximal space and is in good harmony with the adjacent palillae; 4 - the papilla is hyperplastic and covers too much of the implant restoration and/or the adjacent tooth
Time Frame: value changes between examination carried out 3 and 9 months post-op
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group With Implants
Number analyzed (Participants) | 30
score on a scale
  Mesial papilla | 1 [0 to 2]
  Distal papilla | 1 [0 to 2]
Statistical Analysis 1: Comparison: Group With Implants; Test type: Other; p = 0.0005, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.25
Statistical Analysis 2: Comparison: Group With Implants; Test type: Other; p = 0.0034, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1

3. Secondary Outcome: Cone Beam Computed Tomography Examination Taken Right After Implant Installation.
Description: Distance between implant collar and bone margin at buccal and palatal aspect of the crest evaluated on Cone Beam Computed Tomography examination (Pax-i3D Green; Vatech, South Korea).
  The change was calculated from two time points as the value at 12 months minus value at baseline.
Time Frame: Assessed immediately after implantation and 12 months post-op
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group With Implants
Number analyzed (Participants) | 30
mm | 1.99 (1.05)
Statistical Analysis 1: Comparison: Group With Implants; Test type: Other; p = 0.39, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: The definition of adverse event and/or serious adverse event didn't differ from the clinicaltrials.gov.
Arm/Group | Group With Implants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT04243421/Prot_SAP_001.pdf